CLINICAL TRIAL: NCT07121504
Title: Effect of Hybrid Closed-Loop Insulin Delivery System on Glycemic Management in Perioperative Patients With Type 2 Diabetes Receiving Parenteral Nutrition: An Open-Label, Randomized Controlled Trial
Brief Title: Hybrid Closed-Loop for Perioperative Glycemic Control in T2DM With Parenteral Nutrition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Xia Li, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCL-T2D 2025
Record Dates: First submitted 2025-05-22; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: hybrid closed-loop; perioperative; parenteral nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperphagia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid closed-loop insulin delivery system (Experimental): T2DM patients in the experimental group will receive the hybrid closed-loop insulin delivery system.
  Interventions: Device: Hybrid closed-loop insulin delivery system
- Conventional insulin pump with CGM (Active Comparator): T2DM patients in the control group will receive conventional insulin pump therapy with CGM.
  Interventions: Device: conventional insulin pumps combined with CGM

INTERVENTIONS:
Device: Hybrid closed-loop insulin delivery system — Perioperative patients with T2D receiving parenteral nutrition will receive hybrid closed-loop insulin delivery system for glycemic management.
  Arms: Hybrid closed-loop insulin delivery system
Device: conventional insulin pumps combined with CGM — Perioperative patients with T2D receiving parenteral nutrition will receive conventional insulin pumps combined with CGM for glycemic management.
  Arms: Conventional insulin pump with CGM

SUMMARY:
Glycemic control in surgical patients with type 2 diabetes mellitus (T2DM) receiving parenteral nutrition represents a major clinical challenge. This randomized controlled trial evaluates the comparative effectiveness and safety of hybrid closed-loop (HCL) insulin delivery versus conventional insulin pumps combined with continuous glucose monitoring (CGM) in perioperative T2DM patients requiring short-term parenteral nutrition.

DETAILED DESCRIPTION:
This study is a single-center, open-label, 1:1 randomized controlled exploratory trial. Participants were randomly allocated via complete randomization into two groups: the experimental group (hybrid closed-loop insulin delivery system) and the control group (using identical hardware devices, with the experimental group operating in closed-loop mode while the control group in open-loop mode). The intervention duration ranged from 5 to 7 days, adjusted based on glycemic control status, aiming to compare the efficacy and clinical benefits of hybrid closed-loop insulin delivery versus insulin pumps combined with CGM for glycemic management.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Diagnosis of T2DM requiring surgical procedures (duration ≥2 hours) with anticipated short-term total parenteral nutrition (TPN) during the perioperative period (expected hospitalization >72 hours).
3. Glycemic control criteria (meeting any of the following):

   ①HbA1c ≥7.5% or random plasma glucose ≥13.9 mmol/L
   * Established T2DM with poor glycemic control (HbA1c ≥7.5%) despite combination therapy (≥2 oral antidiabetic drugs) ③Insulin-treated patients with suboptimal control (HbA1c ≥7.0%) after adequate dose adjustment.
4. Willing to sign the informed consent form.

Exclusion Criteria:

1. Patients with acute diabetic complications, including: diabetic ketoacidosis (DKA), hyperglycemic hyperosmolar state (HHS), etc.
2. Patients with type 1 diabetes or other specific types of diabetes.
3. Patients with severe organ dysfunction, defined as:

   * Cardiac function ≥Class III (NYHA classification)

     * ALT/AST >3× upper limit of normal (ULN) ③ eGFR ≤30 mL/min/1.73 m²

       * Hemoglobin <90 g/L ⑤ WBC count <4.0×10⁹/L or platelets <90×10⁹/L ⑥ Hemodynamic instability
4. Patients with endocrine disorders affecting glucose metabolism, such as: hyperthyroidism, hypothyroidism, Cushing's syndrome, etc.
5. Patients with known hypersensitivity to any drugs or materials used in the study protocol.
6. Patients who have contraindications to conventional insulin pump therapy.
7. Patients with dermatological conditions (e.g., skin rash, prurigo) or coagulation disorders.
8. Patients with impaired consciousness or psychiatric disorders affecting decision-making capacity or communication ability.
9. Patients who have other conditions deemed unsuitable for trial participation by investigators.
10. Patients who suffer severe surgical complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
CGM-measured Time in Range (TIR 5.6-10.0 mmol/L) | Up to 28 days
  The difference in percentage of time spent within target glucose range (5.6-10.0 mmol/L) between groups, as continuously monitored by a CGM device, to evaluate the effectiveness of hybrid closed-loop insulin delivery versus control in improving glycemic control for perioperative T2DM patients receiving parenteral nutrition.

SECONDARY OUTCOMES:
Time above range (TAR) >10.0 mmol/L | Up to 28 days
  The difference in the CGM-measured percentage of time with sensor glucose values > 10.0 mmol/L between group
Time above range (TAR) >20.0 mmol/L | Up to 28 days
  The difference in the CGM-measured percentage of time with sensor glucose values > 20.0 mmol/L between group
Time below range (TBR) <5.6 mmol/L | Up to 28 days
  The difference in the CGM-measured percentage of time with sensor glucose values <5.6 mmol/L between groups
Time below range (TBR) < 3.9 mmol/L | Up to 28 days
  The difference in the CGM-measured percentage of time with sensor glucose values <3.9 mmol/L between groups
Time below range (TBR) < 3.0 mmol/L | Up to 28 days
  The difference in the CGM-measured percentage of time with sensor glucose values <3.0 mmol/L between groups
Time below range (TBR) < 2.8 mmol/L | Up to 28 days
  The difference in the CGM-measured percentage of time with sensor glucose values <2.8 mmol/L between groups
CGM-measured Mean Glucose Level | Up to 28 days
  CGM-measured mean glucose level between groups
CGM-measured Glucose Standard Deviation (SD) | Up to 28 days
  The difference in the CGM-measured glucose standard deviation between groups. Standard Deviation represents how much glucose levels fluctuate over time from a given average.
CGM-Measured Glucose Coefficient of Variation (CV) | Up to 28 days
  The difference in the CGM-measured glucose coefficient of variation (CV) between groups. The CV is calculated as the ratio of the standard deviation to the mean glucose values for each participant, derived from CGM data.
CGM-Measured Glucose Risk Index (GRI) | Up to 28 days
  The CGM-measured glucose risk index (GRI) between groups. GRI is a comprehensive metric derived from CGM data, designed to quantify the overall risk associated with blood glucose variability. It integrates multiple aspects of glucose levels, including the frequency and severity of both hypo- and hyperglycemic events, as well as the duration of time spent outside the target glucose range.
Insulin dose | Up to 28 days
  The difference in the insulin dose between groups
Preoperative optimization duration (days) | Up to 28 days
  The difference in the preoperative optimization duration between groups
Time in range (TIR) 4.4-10.0 mmol/L | Up to 28 days
  The difference in percentage of time spent within target glucose range (4.4-10.0 mmol/L) between groups, as continuously monitored by a CGM device, to evaluate the effectiveness of hybrid closed-loop insulin delivery versus control in improving glycemic control for perioperative T2DM patients receiving parenteral nutrition.

OTHER OUTCOMES:
Safety outcomes | Up to 28 days
  Safety outcomes will include the difference in the incidence rates of: (1) perioperative infections, (2) hypoglycemia (Level 1: <3.9 mmol/L; Level 2: <3.0 mmol/L; severe: requiring assistance), (3) diabetic ketoacidosis/ketosis, (4) adverse events and device-related adverse events, and (5) all serious adverse events (SAEs), between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Li, MD, PhD, Principal Investigator — Second Xiangya Hospial of Central South University
Locations (1):
- Department of Metabolism and Endocrinology, Second Xiangya Hospital of Centra South University, Changsha, Hunan 410011, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT07121504/SAP_000.pdf